CLINICAL TRIAL: NCT06344559
Title: Theta-burst Stimulation Modulates Criticality and Cognitive Control
Brief Title: Brain Criticality, Oculomotor Control, and Cognitive Effort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Andrew Westbrook, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023001006
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The study will involve three sessions of within-subject, crossover, double-blind transcranial magnetic stimulation with either 1) active intermittent theta burst stimulation, 2) active continuous theta burst stimulation or 3) sham intermittent or continuous theta burst stimulation.
Who Masked: Participant, Investigator
Masking Description: Participants numbers will be assigned three blinded codes which are linked with either sham, active continuous, or active intermittent theta burst stimulation in the stimulator protocol. The investigator will enter the code to initiate the corresponding stimulator protocol, but will not know which protocol is active.
  Half of participants will be assigned a sham code corresponding to sham continuous theta burst stimulation and half will be assigned a sham code corresponding to sham intermittent theta burst stimulation. So, for any given session, either continuous or intermittent theta burst stimulation will be used, but it will be unclear whether the stimulation is active or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Continuous theta burst stimulation (Active Comparator): In a cross-over design, all participants will, in one session, receive continuous theta burst stimulation, to the right frontal eye field. Session order will be counter-balanced across participants, and stimulation protocol will be blinded to participants and the Investigator until after data collection is complete.
  Interventions: Device: transcranial magnetic stimulation
- Intermittent theta burst stimulation (Active Comparator): In a cross-over design, all participants will, in one session, receive intermittent theta burst stimulation, to the right frontal eye field. Session order will be counter-balanced across participants, and stimulation protocol will be blinded to participants and the Investigator until after data collection is complete.
  Interventions: Device: transcranial magnetic stimulation
- Sham theta burst stimulation (Sham Comparator): In a cross-over design, all participants will, in one session, receive sham theta burst stimulation, to the right frontal eye field. Session order will be counter-balanced across participants, and stimulation protocol will be blinded to participants and the Investigator until after data collection is complete.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — The study intervention involves modulation of cortical excitation to inhibition (E/I) balance in the right frontal eye field (FEF) by means of 2 trains of spaced continuous or intermittent theta burst stimulation (cTBS, iTBS, respectively) using a transcranial magnetic stimulation device. The endpoint of this stimulation will be a decrease (cTBS) or increase (iTBS) in the local E/I ratio that should last at least 60 minutes post-stimulation (Chung et al., 2016).
  In separate sessions, all participants will receive either active or stimulation to the FEF. The Investigators will contrast the effects of both iTBS and cTBS to sham stimulation and to each other.

SUMMARY:
The project examines electroencephalography, MRI, and behavioral measures indexing flexibility (critical state dynamics) in the brain when healthy young adults do demanding cognitive tasks, and in response to transcranial magnetic stimulation.

DETAILED DESCRIPTION:
The healthy human brain is a complex, dynamical system which is hypothesized to operate, at rest, near a phase transition - at the boundary between order and chaos. Proximity to this critical point is functionally adaptive as it affords maximal flexibility, dynamic range, and information transmission capacity, with implications for short term memory and cognitive control. Divergence from this critical point has become correlated with diverse forms of psychopathology and neuropathy suggesting that distance from a critical point is both a potential biomarker of disorder and also a target for intervention in disordered brains. The Investigators have further hypothesized that task performance depends on how closely brains operate to criticality during task performance and also that subjective cognitive effort is a reflection of divergence from criticality, induced by engagement with demanding tasks.

A key control parameter determining distance from criticality in a resting brain is hypothesized to be the balance of cortical excitation to inhibition (the "E/I balance"). Transcranial magnetic stimulation is a widely used experimental and clinical tool for neuromodulation and theta-burst stimulation (TBS) protocols are thought to modulate the E/I balance. Here the Investigators test whether cortical dynamics can be systematically modulated away from the critical point with continuous theta-burst stimulation (cTBS) and intermittent theta-burst stimulation (iTBS), which is thought to decrease and increase E/I balance, respectively. Depending on baseline E/I balance prior to stimulation, this will make people's brains either operate closer to, or farther away from critiality and thereby impact on cognitive control and subjective cognitive effort during performance of control-demanding tasks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study and availability for the duration of the study
3. Males and females; Ages 18-45
4. Healthy, neurologically normal with no diagnosed mental or physical illness
5. Willingness to adhere to the MRI and two session stimulation protocol
6. Fluent in English
7. Normal or corrected to normal vision
8. At least twelve years of education (high school equivalent)

Exclusion Criteria:

1. Ongoing drug or alcohol abuse
2. Diagnosed psychiatric or mental illness
3. Currently taking psychoactive medication
4. Prior brain injury
5. Metal in body
6. History of seizures or diagnosis of epilepsy
7. Claustrophobia
8. Pregnant or possibly pregnant
9. Younger than 18 or older than 45
10. Use of medications which potentially lower the usage threshold

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Critical dynamics - immediate effects of cTBS versus sham stimulation | Change in correlations recorded during rest, immediately after stimulation, for active versus sham stimulation.
  Long-range temporal correlations quantified by the scaling exponent, which is derived from EEG data, via detrended fluctuation analysis. Scores range from 0.5 (uncorrelated time series) to 1.0 (correlated time series). Lower scores, indicating weaker correlations, are expected following active continuous theta burst stimulation (cTBS) versus sham stimulation. So, the difference score should be negative, indicating weaker long-range temporal correlations as a result of cTBS, immediately after stimulation.
Functional E/I balance - immediate effects of cTBS versus sham stimulation | Change in the functional E/I balance recorded during rest, immediately after stimulation, for active versus sham stimulation.
  The functional E/I ratio, which is derived from a comparison of band-limited amplitude to the fluctuation function, reflects the balance of excitation versus inhibition driving the associated oscillations. Scores range from approximately 0.5 to 1.5 with values below 1.0 indicating inhibition dominance and values above 1.0 indicating excitation dominance. Lower scores, indicating more inhibition dominance, are expected following active continuous theta burst stimulation (cTBS) versus sham stimulation. So, the difference score should be negative, indicating a lower E/I balance as a result of cTBS, immediately after stimulation.
Avalanche branching ratio - immediate effects of cTBS versus sham stimulation | Change in the avalanche branching ratio recorded during rest, immediately after stimulation, for active versus sham stimulation.
  The growth rate of neuronal avalanches can be estimated from the clustering of high amplitude events in in electroencephalography (EEG) signal. Faster growing avalanches correspond with tighter clustering of events in time. Scores range from approximately 0.5 to 1.5 with values below 1.0 indicating inhibition dominance and values above 1.0 indicating excitation dominance. Lower scores, indicating more inhibition dominance, are expected following active continuous theta burst stimulation (cTBS) versus sham stimulation. So, the difference score should be negative, indicating a lower E/I balance as a result of cTBS, immediately after stimulation.
Critical dynamics - immediate effects of iTBS versus sham stimulation | Change in correlations recorded during rest, immediately after stimulation, for active versus sham stimulation.
  Long-range temporal correlations quantified by the scaling exponent, which is derived from EEG data, via detrended fluctuation analysis. Scores range from 0.5 (uncorrelated time series) to 1.0 (correlated time series). Higher scores, indicating stronger correlations, are expected following active intermittent theta burst stimulation (iTBS) versus sham stimulation. So, the difference score should be positive, indicating stronger long-range temporal correlations as a result of iTBS, immediately after stimulation.
Functional E/I balance - immediate effects of iTBS versus sham stimulation | Change in the functional E/I balance recorded during rest, immediately after stimulation, for active versus sham stimulation.
  The functional E/I ratio, which is derived from a comparison of band-limited amplitude to the fluctuation function, reflects the balance of excitation versus inhibition driving the associated oscillations. Scores range from approximately 0.5 to 1.5 with values below 1.0 indicating inhibition dominance and values above 1.0 indicating excitation dominance. Higher scores, indicating more excitation dominance, are expected following active intermittent theta burst stimulation (iTBS) versus sham stimulation. So, the difference score should be positive, indicating a higher E/I balance as a result of iTBS, immediately after stimulation.
Avalanche branching ratio - immediate effects of iTBS versus sham stimulation | Change in the avalanche branching ratio recorded during rest, immediately after stimulation, for active versus sham stimulation.
  The growth rate of neuronal avalanches can be estimated from the clustering of high amplitude events in in electroencephalography (EEG) signal. Faster growing avalanches correspond with tighter clustering of events in time. Scores range from approximately 0.5 to 1.5 with values below 1.0 indicating inhibition dominance and values above 1.0 indicating excitation dominance. Higher scores, indicating more excitation dominance, are expected following active intermittent theta burst stimulation (iTBS) versus sham stimulation. So, the difference score should be positive, indicating a higher E/I balance as a result of iTBS, immediately after stimulation.
Memory-guided saccade accuracy - effects of cTBS versus sham stimulation | Change in degrees of visual angle error estimated 44 minutes after stimulation, for cTBS versus sham stimulation.
  Accuracy on the memory-guided saccade task, as quantified by mean degrees of visual angle deviation typically range from ~1.0 to 5.0 degrees, with higher scores indicating higher inaccuracy. Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. Because criticality implies susceptibility and flexibility, stimulation protocols which make the FEF operate closer to criticality, relative to sham stimulation, will show bigger errors in degrees of visual angle.
Memory-guided saccade accuracy - effects of iTBS versus sham stimulation | Change in degrees of visual angle error estimated 44 minutes after stimulation, for iTBS versus sham stimulation.
  Accuracy on the memory-guided saccade task, as quantified by mean degrees of visual angle deviation typically range from ~1.0 to 5.0 degrees, with higher scores indicating higher inaccuracy. Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. Because criticality implies susceptibility and flexibility, stimulation protocols which make the FEF operate closer to criticality, relative to sham stimulation, will show bigger errors in degrees of visual angle.
Anti-saccade accuracy - effects of cTBS versus sham stimulation | Change in percent accuracy estimated 12 minutes after stimulation, for cTBS versus sham stimulation.
  Accuracy on the anti-saccade task, as quantified by mean percent of correct saccades away from a cue typically ranges between 80% and 100% correct. Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. Because criticality implies greater inter-regional communication between top-down control regions and sensorimotor cortex, stimulation protocols which make the FEF operate closer to criticality, relative to sham stimulation, will a higher perfect increase in accuracy as a result of stimulation.
Anti-saccade accuracy - effects of iTBS versus sham stimulation | Change in percent accuracy estimated 12 minutes after stimulation, for iTBS versus sham stimulation.
  Accuracy on the anti-saccade task, as quantified by mean percent of correct saccades away from a cue typically ranges between 80% and 100% correct. Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. Because criticality implies greater inter-regional communication between top-down control regions and sensorimotor cortex, stimulation protocols which make the FEF operate closer to criticality, relative to sham stimulation, will a higher perfect increase in accuracy as a result of stimulation.
Subjective effort discounting - cTBS versus sham stimulation | Change in subjective value estimated 72 minutes after stimulation, for cTBS versus sham stimulation.
  Subjective values as estimated from an effort discounting procedure as a discounted offer ranging from 0.0 (full effort discounting) to 1.0 (no effort discounting). Lower values indicate that people find subjective effort to be more costly. Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. We hypothesize that divergence from criticality underlies phenomenological effort. So, we predict that stimulation which makes people's brains operate closer to criticality relative to sham will experience less effort and have a higher subjective value.
Subjective effort discounting - iTBS versus sham stimulation | Change in subjective value estimated 72 minutes after stimulation, for iTBS versus sham stimulation.
  Subjective values as estimated from an effort discounting procedure as a discounted offer ranging from 0.0 (full effort discounting) to 1.0 (no effort discounting). Lower values indicate that people find subjective effort to be more costly. Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. We hypothesize that divergence from criticality underlies phenomenological effort. So, we predict that stimulation which makes people's brains operate closer to criticality relative to sham will experience less effort and have a higher subjective value.
Subjective effort rating - cTBS versus sham stimulation | Change in subjective value estimated 70 minutes after stimulation, for cTBS versus sham stimulation.
  Likert ratings of subjective effort randing from 1 (low effort) to 10 (high effort). Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. We hypothesize that divergence from criticality underlies phenomenological effort. So, we predict that stimulation which makes people's brains operate closer to criticality relative to sham will experience less effort and have a higher subjective value.
Subjective effort rating - iTBS versus sham stimulation | Change in subjective value estimated 70 minutes after stimulation, for iTBS versus sham stimulation.
  Likert ratings of subjective effort randing from 1 (low effort) to 10 (high effort). Theta burst stimulation to the FEF should modulate cortical excitability making the FEF in some people's brains operate closer to criticality, and in others' brains, operate farther from criticality. We hypothesize that divergence from criticality underlies phenomenological effort. So, we predict that stimulation which makes people's brains operate closer to criticality relative to sham will experience less effort and have a higher subjective value.

CONTACTS AND LOCATIONS:
Overall Officials: John A Westbrook, PhD, Principal Investigator — Rutgers University
Locations (1):
- Center for Advanced Human Brain Imaging Research, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
All anonymized data will be made publicly available at the conclusion of the trial at Rutgers University's (RUresearch) Data Portal.

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210

DOCUMENTS (2):
  • Study Protocol (2024-03-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT06344559/Prot_000.pdf
  • Informed Consent Form (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT06344559/ICF_001.pdf